CLINICAL TRIAL: NCT02055833
Title: Intensive Nutritional Counseling in Head-neck Cancer Patients Undergoing Radiotherapy: a Randomized, Controlled Trial
Brief Title: Intensive Nutritional Counseling in Head-neck Cancer Patients Undergoing Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Nestlè Health Science (Unknown); Akern Srl (Industry)
Responsible Party: Principal Investigator, Emanuele Cereda, MD, PhD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120001310
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2016-08

CONDITIONS: Head-neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive nutritional counseling (Experimental): Nutritional counseling (follow-up visits once a week for 6 weeks [during radiotherapy] and at 1 month and at 3 months since the end of radiotherapy) + n-3 polyunsaturated fatty acids-enriched oral nutritional supplements (1-2 bottles/day)
  Interventions: Dietary Supplement: Intensive nutritional counseling
- Nutritional counseling (Active Comparator): Nutritional counseling (follow-up visits once a week for 6 weeks [during radiotherapy] and at 1 month and at 3 months since the end of radiotherapy)
  Interventions: Other: Nutritional counseling

INTERVENTIONS:
Dietary Supplement: Intensive nutritional counseling — Intensive nutritional counseling: nutritional counseling + oral nutritional supplements
  Other Names: Resource Support Plus (Nestlè Health Science)
  Arms: Intensive nutritional counseling
Other: Nutritional counseling — Nutritional counseling
  Arms: Nutritional counseling

SUMMARY:
In head-neck cancer patients undergoing radiotherapy (RT) malnutrition is associated with impaired quality of life, reduced survival, more frequent treatment interruptions and dose reductions. The international guidelines recommend early nutritional support in the presence of nutritional risk, as it allows preventing or treating malnutrition and improving the clinical outcomes, as well as the tolerability of oncologic treatments. Previous nutritional intervention trials in head-neck cancer patients have been conducted on small samples and did not clarify the role of oral nutritional supplements (ONS). Accordingly, although current guidelines recommend as grade A the use of ONS associated with dietary counseling for head-neck cancer patients undergoing RT, the efficacy of this nutritional intervention still needs to be evaluated in adequately sized and randomized clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed head-neck cancer
* indication to radiotherapy
* Eastern Cooperative Oncology Group performance status <=2
* availability to planned measurements and to written informed consent.

Exclusion Criteria:

* age <18 years
* ongoing artificial nutrition
* refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2013-09; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Body weight | 6 weeks
  Change in body weight at the end of radiotherapy (after 6 weeks)

SECONDARY OUTCOMES:
Body weight | 3 months
  Change in body weight at 1 month since the end of radiotherapy
Body weight | 5 months
  Change in body weight at 3 months since the end of radiotherapy
Quality of life | 5 months
  Trends in quality of life during the study (assessment: at the end of radiotherapy; at 1 month and at 3 months since the end of radiotherapy)
Handgrip strength | 5 months
  Trends in handgrip strength during the study (assessment: at the end of radiotherapy; at 1 month and at 3 months since the end of radiotherapy)
Phase angle | 5 months
  Trends in phase angle (as surrogate of body composition) during the study (assessment: at the end of radiotherapy; at 1 month and at 3 months since the end of radiotherapy)

OTHER OUTCOMES:
Feasibility of radiotherapy | 6 weeks
  Described as: number of interruptions >5 days; total duration (days); dose reduction

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Cereda, MD, PhD, Principal Investigator — Nutrition and Dietetics Service, Fondazione IRCCS Policlinico San Matteo; Riccardo Caccialanza, MD, Study Director — Nutrition and Dietetics Service, Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Nutrition and Dietetics Service, Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

REFERENCES:
- [Background] Langius JA, Zandbergen MC, Eerenstein SE, van Tulder MW, Leemans CR, Kramer MH, Weijs PJ. Effect of nutritional interventions on nutritional status, quality of life and mortality in patients with head and neck cancer receiving (chemo)radiotherapy: a systematic review. Clin Nutr. 2013 Oct;32(5):671-8. doi: 10.1016/j.clnu.2013.06.012. Epub 2013 Jun 26. PMID 23845384
- [Background] Baldwin C, Spiro A, Ahern R, Emery PW. Oral nutritional interventions in malnourished patients with cancer: a systematic review and meta-analysis. J Natl Cancer Inst. 2012 Mar 7;104(5):371-85. doi: 10.1093/jnci/djr556. Epub 2012 Feb 15. PMID 22345712
- [Background] Arends J, Bodoky G, Bozzetti F, Fearon K, Muscaritoli M, Selga G, van Bokhorst-de van der Schueren MA, von Meyenfeldt M; DGEM (German Society for Nutritional Medicine); Zurcher G, Fietkau R, Aulbert E, Frick B, Holm M, Kneba M, Mestrom HJ, Zander A; ESPEN (European Society for Parenteral and Enteral Nutrition). ESPEN Guidelines on Enteral Nutrition: Non-surgical oncology. Clin Nutr. 2006 Apr;25(2):245-59. doi: 10.1016/j.clnu.2006.01.020. Epub 2006 May 12. PMID 16697500
- [Derived] Martin B, Cereda E, Caccialanza R, Pedrazzoli P, Tarricone R, Ciani O. Cost-effectiveness analysis of oral nutritional supplements with nutritional counselling in head and neck cancer patients undergoing radiotherapy. Cost Eff Resour Alloc. 2021 Jun 15;19(1):35. doi: 10.1186/s12962-021-00291-7. PMID 34130709
- [Derived] Cereda E, Cappello S, Colombo S, Klersy C, Imarisio I, Turri A, Caraccia M, Borioli V, Monaco T, Benazzo M, Pedrazzoli P, Corbella F, Caccialanza R. Nutritional counseling with or without systematic use of oral nutritional supplements in head and neck cancer patients undergoing radiotherapy. Radiother Oncol. 2018 Jan;126(1):81-88. doi: 10.1016/j.radonc.2017.10.015. Epub 2017 Oct 27. PMID 29111172